CLINICAL TRIAL: NCT03440996
Title: Comparison of Clinpro™ 5000 1.1% Sodium Fluoride Anti-Cavity Toothpaste, Clinpro™ Tooth Crème, and MI-Paste Plus for the Prevention and Reduction of White Spot Lesions in Orthodontic Treatment
Brief Title: Comparison of Three Toothpastes for the Prevention and Reduction of White Spot Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Chung How Kau, Professor and Chairman, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1122614
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: White Spot Lesion; Orthodontic Treatment; Decalcification; Teeth
Keywords: toothpaste
MeSH Terms: interventions — Toothpastes; GC dentin cement

STUDY DESIGN:
Intervention Model Description: Three groups of 30 subjects (one group with Clinpro™ 5000, one group with MI-Paste Plus, and one group with Clinpro™ Tooth Crème) each will be evaluated as a protocol for the reduction of white spot lesions at the start of orthodontic treatment. Subjects will be recruited through the Orthodontic Postgraduate Clinic at the University of Alabama at Birmingham School of Dentistry.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Clinpro™ 5000 (Experimental): Participants will use Clinpro™ 5000 to brush their teeth for two minutes twice daily for 4 months.
  Interventions: Other: Clinpro™ 5000
- Clinpro™ Tooth Crème (Experimental): Participants will use Clinpro™ Tooth Crème to brush their teeth for two minutes twice daily for 4 months.
  Interventions: Other: Clinpro™ Tooth Crème
- MI-Paste Plus (Active Comparator): Participants will use MI-Paste Plus to brush their teeth for two minutes twice daily for 4 months.
  Interventions: Other: MI-Paste Plus

INTERVENTIONS:
Other: Clinpro™ 5000 — Clinpro™ 5000 with 1.1% Sodium Fluoride is a new anti-cavity toothpaste, and is currently available and have been shown in some initial case reports to be useful in the reduction of white spot lesions. Clinpro™ restores minerals and helps you produce saliva. The Clinpro™ products are advanced formulas containing an innovative tri-calcium phosphate ingredient. It is available exclusively from 3M ESPE. Clinpro™ contains fluoride as well as calcium and phosphate, which are components naturally found in saliva.
  Other Names: Toothpaste produced by 3M ESPE.
  Arms: Clinpro™ 5000
Other: Clinpro™ Tooth Crème — Clinpro™ Tooth Crème with 0.21% Sodium Fluoride is a new anti-cavity toothpaste, and is currently available and have been shown in some initial case reports to be useful in the reduction of white spot lesions. Clinpro™ restores minerals and helps you produce saliva. The Clinpro™ products are advanced formulas containing an innovative tri-calcium phosphate ingredient. It is available exclusively from 3M ESPE. Clinpro™ contains fluoride as well as calcium and phosphate, which are components naturally found in saliva.
  Other Names: Toothpaste produced by 3M ESPE.
  Arms: Clinpro™ Tooth Crème
Other: MI-Paste Plus — MI-Paste Plus is a widely used anti-cavity toothpaste on the market and it is used as a control group in this study.
  Other Names: Toothpaste produced by GC America
  Arms: MI-Paste Plus

SUMMARY:
The purpose of the study is to determine if Clinpro™ 5000, Clinpro™ Tooth Crème, or MI-Paste Plus has an effect on the formation and resolution of white spot lesions for patients undergoing orthodontic treatment. This study will include 90 patients in the UAB Orthodontic Clinic.

DETAILED DESCRIPTION:
During the course of orthodontic treatment, the practitioner normally faces two common iatrogenic treatment side effects: root resorption and enamel decalcification, with the latter occurring at a much higher frequency. While the processes that lead to enamel demineralization are understood, methods to diminish or perhaps eliminate degradation of enamel surfaces are being searched for. Several approaches have been formulated to counteract demineralization of tooth structure. One approach involves patient compliance and consists of in-depth oral hygiene instructions, in-office fluoride applications, and at-home fluoride rinses, gels, and varnishes. An alternative approach, which possesses potential benefit regardless of patient compliance, includes the use of fluoride-releasing agents, such as composites, glass ionomers, sealants, and elastomeric ties.

Enamel decalcification or white spot formation, is a phenomenon occurring primarily on smooth enamel surfaces of teeth, notably within the gingival third of the crown. Demineralized enamel, the precursor to caries formation, can be attributed to fixed orthodontic appliances, and prolonged exposure to bacterial plaque. Bacterial plaque promotes the accumulation of acidic byproducts and demineralization that leads to successive changes in the optical properties of subsurface demineralized enamel. Progression to clinically detectable white spot lesions may occur as early as one month following the placement of orthodontic appliances.

Two new anti-cavity toothpastes, Clinpro™ 5000 with 1.1% Sodium Fluoride and Clinpro™ Tooth Crème with 0.21% Sodium Fluoride, are currently available and have been shown in some initial case reports to be useful in the reduction of white spot lesions. Clinpro™ restores minerals and helps you produce saliva. Both the Clinpro™ products are advanced formulas containing an innovative tri-calcium phosphate ingredient. They are available exclusively from 3M ESPE. Clinpro™ contains fluoride as well as calcium and phosphate, which are components naturally found in saliva.

Thus, this study will compare Clinpro™ 5000 1.1% Sodium Fluoride Anti-Cavity Toothpaste, Clinpro™ Tooth Crème, and MI-Paste Plus for the prevention and reduction of white spot lesions during orthodontic treatment.

ELIGIBILITY:
INCLUSION CRITERIA

1. Permanent dentition
2. Patients that in the opinion of the investigator will be compliant with the use of the paste
3. Patients who have not used extensive fluoride regimes
4. 12 years and older
5. Subjects must use a non-fluoridated toothpaste (such as Tom's of Maine) for a one-week period prior to starting this trial.

EXCLUSION CRITERIA

1. Any medical or dental condition that in the opinion of the investigator could impact study results during the expected length of the study.
2. Patient is currently using any investigational drug.
3. Patient plans to relocate or move within six months of enrollment.
4. Patients who have or are currently undergoing fluoride treatment for white spot lesions.
5. Patients with IgE Casein Allergy

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2011-01-14 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-12-30 (Actual)

PRIMARY OUTCOMES:
Photographic records and clinical examination | Subjects will be reviewed every 4 weeks. Photographs will be taken for 4 times at monthly intervals. Changes will be compared and assessed. The duration of the observation is an average of 4 months.
  Photographic records will be used to determine the improvements in the white spot lesions. A standard intra-oral photographic camera will be utilized and the photographs will be taken in a light controlled environment and photographs will be captured in a pre-set photographic protocol. The Enamel decalcification index (EDI) will be used to determine the number of white spot lesions present at each time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Chung H Kau, BDS, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Kau CH, Wang J, Palombini A, Abou-Kheir N, Christou T. Effect of fluoride dentifrices on white spot lesions during orthodontic treatment: A randomized trial. Angle Orthod. 2019 May;89(3):365-371. doi: 10.2319/051818-371.1. Epub 2019 Feb 5. PMID 30719933

DOCUMENTS (2):
  • Study Protocol (2011-02-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT03440996/Prot_000.pdf
  • Statistical Analysis Plan (2011-02-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT03440996/SAP_001.pdf